CLINICAL TRIAL: NCT05280743
Title: Avoiding Adverse Opioid Outcomes With Proactive Precision Care Following Cesarean Delivery
Brief Title: Precision Opioid Care After Cesarean Delivery (PRECISE-CD)
Acronym: PRECISE-CD
Status: Completed | Type: Observational
Sponsor: Grace Lim, MD, MS (Other)
Responsible Party: Sponsor-Investigator, Grace Lim, MD, MS, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: STUDY21070164
Record Dates: First submitted 2022-03-06; First posted 2022-03-15 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Cesarean Section Complications; Opioid Use
Keywords: Personalized Care
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pharmacogenetic (PG) Blood Samples: A blood sample will be collected to assess polymorphisms of genotypes, epigenetics, and gene expression affecting opioid effectiveness, metabolism and transport. CYP2D6 genotyping will be utilized to characterize CYP2D6 Poor Metabolizers (PMs) and Ultrarapid Metabolizers (UMS). Polymorphisms of OPRM1, COMT, and GCH1 have been associated with intensity and chronicity of post-surgical pain. The Illumina Human Omni5M+exome GWAS array (4.3 million SNPs) or equivalent GWAS panel will help us explore additional genetic variants while allowing unbiased exploration of additional154 biologically relevant genetic variants cost-effectively in all study participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MATERNAL cohort: Nursing mothers who underwent Cesarean Delivery and who are receiving oxycodone to treat post-operative pain
  Interventions: Drug: Oxycodone
- NEONATE-INFANT cohort: Neonate" encompasses a newborn from the age of birth until <28 days of life. "Infant" refers to the period of 28 days of life until 1 year of life.
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Oxycodone — exposure to opioids after Cesarean Section
  Other Names: Opioid Exposure

SUMMARY:
The purpose of this research is to study serious clinical problems from surgical pain and the use of oxycodone or other opioids in women having a Cesarean Delivery to improve the safety and efficacy of surgical pain relief. This research will ultimately improve the safety and efficacy of surgical pain relief with opioids by preoperative risk predictions and personalized care with the right dose of the right analgesic for each patient.

DETAILED DESCRIPTION:
The overall objective is to determine the impact of risk factors on oxycodone and other opioid's adverse postoperative outcomes and to personalize dosing in women having a Cesarean Delivery. For the purpose of this study, immediate adverse postoperative outcomes are characterized as Respiratory Depression (RD), Postoperative Nausea and Vomiting (PONV), and inadequate surgical pain relief. Long-term adverse postoperative outcomes are characterized as Chronic Persistent Surgical Pain (CPSP) and Opioid Dependence (OD).

The central hypothesis is that specific genetic factors in pain-opioid pathways significantly impact oxycodone and opioid dosing, analgesia, immediate adverse effects (RD and PONV), and long-term adverse outcomes (CPSP and OD).

The aims of this project are to validate genetic variants and to develop a test for preoperative risk prediction in lactating mothers and breastfed babies following cesarean delivery (CD). There is an urgent and unmet critical need for reliable technology to improve safety and effectiveness of opioid use in special populations.

Aim 1. Validate and identify genetic risk factors associated with postoperative opioid adverse effects, PONV and RD in adult nursing mothers following CD.

Investigators hypothesize that with standardized and genotype-blinded perioperative care, specific variants will identify nursing mothers at risk for opioid-induced RD and PONV (primary outcome), OD and severe pain following CD. In addition, genetic variants will identify risk for opioid-induced sedation and adverse effects in breastfed infants. In addition to clinical outcomes, the investigators will collect post-CD cost of care including length of stay.

Aim 2. Develop a laboratory-developed test (LDT) at University of Pittsburgh Genome Center (UGC) for preoperative genetic risk prediction and decision support for surgical patients to prevent adverse opioid outcomes. Investigators will develop a minimum viable product (MVP) (CPT code: 81227), a refined multi-gene panel in UGC's CLIA certified laboratory with a robust combinatorial pharmacogenetic decision support to personalize surgical analgesia with precise opioid use in children and adults, and to prevent RD, PONV, CPSP and OD.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Adult women (>18 y) and their infants
* All races
* ASA physical status 2 to 3
* Cesarean delivery at UPMC Magee
* Planned breast feeding mothers and their infants

Exclusion Criteria:

* Serious illnesses or condition of either mother or infant precluding ability to participate in study procedures
* Multiple gestation pregnancies
* Preoperative severe pain and opioid use/misuse
* Allergy to oxycodone
* Women with opioid use disorder
* Any known condition that anticipates neonatal observation in NICU immediately after birth
* General anesthesia anticipated or converted intraoperatively
* Expected non-viable current gestation or serious neonatal health comorbidities anticipated prior to delivery
* Severe neurological disorder: any known untreated or uncontrolled seizure disorder, pre-eclampsia with severe features, pre-eclampsia requiring magnesium, elevated ICP other than benign intracranial hypertension condition, or conditions at the discretion of PI
* Liver disease: any known abnormal live function tests, or conditions at the discretion of PI
* Renal diseases: any chronic or acute renal insufficiency, or pre-eclampsia diagnosis with abnormal renal function i.e.: severe features, or conditions at the discretion of PI.
* Contraindications to neuraxial anesthesia, neuraxial morphine, acetaminophen, or NSAIDs which are standard parts of post-cesarean multimodal analgesia

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Participants who have Cesarean Delivery and who plan to breast feed their infants
Sampling Method: Non-Probability Sample
Enrollment: 341 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-09-24 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Opioid-Induced Adverse Effects-PROPORTION of maternal participants with RD | From time of surgery to time of discharge up to 3 days post-surgery
  Respiratory depression (RD) measured as Yes or No in occurrence.
Opioid-Induced Adverse Effects-PROPORTION of maternal participants with PONV | From time of surgery to time of discharge up to 3 days post-surgery
  Postoperative Nausea and Vomiting (PONV) Intensity Scale. Participants will be categorized as Clinically relevant (Yes) or Not clinically relevant (No) Nausea and Vomiting from the PONV scale. Clinically important PONV is defined as a total score >50 at any time throughout the study period.

SECONDARY OUTCOMES:
Maternal Post-operative Pain Scores | From time of delivery to 12-month post-surgery
  Numerical Rating Scale (NRS). The pain scale is from 0 to 10, 0 being "no pain" and 10 being "the worst pain imaginable"
Total Maternal Inpatient Opioid Use | From time of surgery to discharge-- up to 3 days post-surgery
  measured in milligrams of Morphine Equivalents
Extended Hospital Length of Stay-Maternal | From surgery to 72 hours postoperation
  Yes/No Proportion of Women discharged beyond 72-hours post-surgery
Length of prescribed opioid use (For Mothers; in days) | From day of surgery to 12-month post-surgery
  Number of days patients take opioids post-surgery.
Neonatal Sedation-- PROPORTION of infants with Sedation | From birth to 7-days post-birth
  Defined as YES (any sleeping > 4 hours in hospital or first week of life) or NO (sleeping) less than 4 hours at a time.
Neonatal Respiratory Depression--PROPORTION of neonates diagnosed with RD | From birth to time of discharge (up to 3 days post-birth)
  Yes/No Yes: Defined as respiratory rate 8 or fewer breaths per minute
Extended Hospital Length of Stay-Neonate | From time of delivery to 72-hours post-delivery
  Yes/No Proportion of neonates staying in hospital longer than 72-hours (Yes)
Neonatal Limpness (reporting limpness > 0, or not limp =0) | From birth to 72-hours post-delivery
  Proportion of Infants with Limpness reported
Proportion of Neonates Exhibiting opioid withdrawal | Birth to 3-days postpartum (or discharge from hospital)
  SOWSS Sophia Observation Withdrawal Symptoms-Scale; Yes (withdrawal symptoms (scores >4)/No (withdrawal symptoms < 4)

CONTACTS AND LOCATIONS:
Overall Officials: Grace Lim, MD MSc, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee Women's Hospital of UPMC, Pittsburgh, Pennsylvania, United States